CLINICAL TRIAL: NCT00002084
Title: A Comparative Trial of Valacyclovir Hydrochloride ( 256U87 ) and Acyclovir for the Suppression of Anogenital Herpes Infections in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 104B; 07
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Herpes Simplex; HIV Infections
Keywords: Acyclovir; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Anus Diseases; Herpes Genitalis
MeSH Terms: conditions — Herpes Simplex; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Anus Diseases; Herpes Genitalis | interventions — Valacyclovir; Acyclovir

INTERVENTIONS:
Drug: Valacyclovir hydrochloride
Drug: Acyclovir

SUMMARY:
To determine the safety and efficacy of oral valacyclovir hydrochloride ( 256U87 ) compared to acyclovir in the treatment of recurrent anogenital herpes in HIV-infected patients with CD4 counts = or > 100 cells/mm3.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection with CD4 counts = or > 100 cells/mm3.
* Documented culture of anogenital herpes simplex virus (HSV) within the last 5 years.
* History of recurrent anogenital HSV infection, with a recurrence (with or without culture) within 1 year prior to study.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Malabsorption or vomiting that would potentially limit the retention and absorption of oral therapy.

Concurrent Medication:

Excluded:

* Systemic antiherpes medication.
* Interferon.

Patients with the following prior conditions are excluded:

History of hypersensitivity to acyclovir.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (46):
- United States (46):
  - Univ of South Alabama, Mobile, Alabama
  - Univ of Arizona / Health Science Ctr, Tucson, Arizona
  - Combat Group, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Infectious Disease Med Group / Adult Immunology Clinic, Oakland, California
  - UCI Med Ctr, Orange, California
  - UCSD Med Ctr, San Diego, California
  - San Diego Naval Hosp, San Diego, California
  - ViRx Inc, San Francisco, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Dr Marcus Conant, San Francisco, California
  - West Haven Veterans Administration Med Ctr, West Haven, Connecticut
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Whitman - Walker Clinic, Washington D.C., District of Columbia
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Veterans Administration Med Ctr / Regional AIDS Program, Washington D.C., District of Columbia
  - Univ of South Florida, St. Petersburg, Florida
  - Emory Univ School of Medicine, Atlanta, Georgia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Northwestern Memorial Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Infectious Diseases Research Clinic / Indiana Univ Hosp, Indianapolis, Indiana
  - Univ of Iowa Hosp & Clinic, Iowa City, Iowa
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - Univ of Maryland at Baltimore, Baltimore, Maryland
  - St Paul Ramsey Med Ctr, Saint Paul, Minnesota
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - Univ of Missouri at Kansas City School of Medicine, Kansas City, Missouri
  - St Louis Univ, St Louis, Missouri
  - Beth Israel Med Ctr, New York, New York
  - Saint Vincent's Hosp and Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Univ of Pittsburgh / Graduate School of Public Health, Pittsburgh, Pennsylvania
  - Roger Williams Med Ctr, Providence, Rhode Island
  - Regional Med Ctr at Memphis, Memphis, Tennessee
  - Dallas Associated Dermatologists, Dallas, Texas
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Thomas Audetta Clinic, Houston, Texas
  - Baylor College of Medicine / Texas Med Ctr, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - MacGregor Med Association, Houston, Texas
  - Univ TX Med Branch / Ctr for Clinical Studies, Nassau Bay, Texas
  - Med College of Virginia, Richmond, Virginia